CLINICAL TRIAL: NCT04864951
Title: HPV Prevalence in Transpersons - a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophie Pils (Other)
Responsible Party: Sponsor-Investigator, Sophie Pils, Clinical Professor, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1186/2021
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Papillomavirus Infection; Transsexualism
MeSH Terms: conditions — Papillomavirus Infections; Transsexualism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transpeople (Other): 1x urine sampling for HPV analysis
  1x survey
  Interventions: Diagnostic Test: Colli-Pee urine collection device; Other: Survey

INTERVENTIONS:
Diagnostic Test: Colli-Pee urine collection device — first-void urine is collected using Colli-Pee and subsequently analyzed using Anyplex™ II HPV HR Detection from Seegene.
Other: Survey — Subjects are asked to complete a survey that includes questions about sexual orientation, hormone therapy, gender reassignment surgery, number of sexual partners, HPV vaccination, and smoking

SUMMARY:
In this study, Human Papilloma Virus (HPV) prevalence will be determined once in the urine of 200 trans people. In addition, subjects will be asked to complete a questionnaire about their sexual orientation, which is adapted from the largest published study.

DETAILED DESCRIPTION:
All transpeople who visit the outpatient clinic are asked to participate in the study. After being informed and signing the Informed Consent Form, the subjects are asked to give first-void urine and fill out the survey. The urine samples are sent pseudonymously to the University of Ljubljana for analysis. The subjects will be informed about their results within 3 weeks.If the result is positive, the subjects will be offered voluntary further care in our HPV outpatient clinic. However, this will take place outside the study. The data collected there can be used for further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Transpeople
* Age over 18 years
* Sufficient knowledge of German

Exclusion Criteria:

* Age under 18 years
* Insufficient knowledge of German

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — all study participants classify themselves as transmen, transwomen, genderqueer, non-binary or other gender identity
Enrollment: 203 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
HPV prevalence in transpeople | one year
  HPV prevalence in transpeople

CONTACTS AND LOCATIONS:
Overall Officials: Elmar Joura, MD, Principal Investigator — Medical University of Vienna, Department of Obstetrics and Gynecology
Locations (2):
- Medical University of Vienna, Vienna, Austria
- Institute of Microbiology and Immunology Faculty of Medicine, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reisner SL, Deutsch MB, Peitzmeier SM, White Hughto JM, Cavanaugh TP, Pardee DJ, McLean SA, Panther LA, Gelman M, Mimiaga MJ, Potter JE. Test performance and acceptability of self- versus provider-collected swabs for high-risk HPV DNA testing in female-to-male trans masculine patients. PLoS One. 2018 Mar 14;13(3):e0190172. doi: 10.1371/journal.pone.0190172. eCollection 2018. PMID 29538411
- [Derived] Pils S, Mlakar J, Poljak M, Domjanic GG, Kaufmann U, Springer S, Salat A, Langthaler E, Joura EA. HPV screening in the urine of transpeople - A prevalence study. EClinicalMedicine. 2022 Oct 12;54:101702. doi: 10.1016/j.eclinm.2022.101702. eCollection 2022 Dec. PMID 36263396